CLINICAL TRIAL: NCT05459428
Title: Artificial Intelligence Confocal Laser Endomicroscopy for Real-time Assessment of Gastric Cancer Risk: a Prospective Exploratory Study
Brief Title: Artificial Intelligence Confocal Laser Endomicroscopy for Real-time Assessment of Gastric Cancer Risk.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Other Study IDs: 2022-SDU-QILU-108
Record Dates: First submitted 2022-07-08; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Intestinal Metaplasia of Gastric Mucosa; Confocal Laser Endomicroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — When a gastric mucosal lesion is found using confocal laser microendoscopy, endoscopist will take biopsy for histology examination. In addition, random biopsies to ensure at least four biopsies from the gastric antrum and body to cauculate the OLGIM
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confocal laser endomicroscopy scoring of the extent of intestinal metaplasia: Get pictures and Videos from gastric antrum body and angle by confocal laser endomicroscopy in order to calculate the CGGIM score.
- Artificial intelligence scoring of the extent of intestinal metaplasia: Get pictures and Videos from gastric antrum body and angle by Artificial intelligence in order to calculate the CGGIM score.

SUMMARY:
Current national guidelines recommend the use of OLGIM score to evaluate the risk of gastric cancer in patients, and close gastroscopic monitoring should be performed after OLGIM grade III/IV. However, it would not be clinically feasible to require at least four biopsies. Confocal laser endomicroscopy is able to magnify the tissue by 1000X, which can be seen at the cellular level. Observing goblet cells under Confocal laser endomicroscopy is simpler and diagnostic accuracy is comparable to pathology. Confocal laser endomicroscopy enables better assessment of intestinal metaplasia in gastric mucosa, thus quantifying the risk of gastric cancer and avoiding multiple biopsies.

DETAILED DESCRIPTION:
Globally, gastric cancer is the fifth most prevalent malignancy and the third leading cause of cancer mortality. Current national guidelines recommend the use of OLGIM score to evaluate the risk of gastric cancer in patients, and close gastroscopic monitoring should be performed after OLGIM grade III/IV. However, it would not be clinically feasible to require at least four biopsies. Confocal laser endomicroscopy is able to magnify the tissue by 1000X, which can be seen at the cellular level. Observing goblet cells under Confocal laser endomicroscopy is simpler and diagnostic accuracy is comparable to pathology. Confocal laser endomicroscopy enables better assessment of intestinal metaplasia in gastric mucosa, thus quantifying the risk of gastric cancer and avoiding multiple biopsies. The investigators aim to design the CGGIM scores to evaluate gastric cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-80 years undergoing the confocal laser endomicroscopy examination

Exclusion Criteria:

* Patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric disorders who cannot participate in gastroscopy
* Patients with previous surgical procedures on the stomach
* Patients with contraindications to biopsy
* Patients who refuse to sign the informed consent form

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People at high risk of developing stomach cancer
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Endoscopists concluded the sensitivity of CGGIM score in the diagnosis of OLGIM III/IV | 2 years
  The confocal grading of gastric intestinal metaplasia (CGGIM) may be used to assess a patient's risk by the endoscopic assessment of IM in the antrum, incisura, and corpus with the use of confocal laser endomicroscopy. The minimum score is 0 and the maximum score is 10. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients. CGGIM scores were calculated to be compared with OLGIM based on the results of the endoscopist 's procedure.
Endoscopists derive the specificity of CGGIM score in the diagnosis of OLGIM III/IV | 2 years
  The confocal grading of gastric intestinal metaplasia (CGGIM) may be used to assess a patient's risk by the endoscopic assessment of IM in the antrum, incisura, and corpus with the use of confocal laser endomicroscopy. The minimum score is 0 and the maximum score is 10. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients. CGGIM scores were calculated to be compared with OLGIM based on the results of the endoscopist 's procedure.
Accuracy of CGGIM Score for Diagnosing OLGIM III/IV by Endoscopists | 2 years
  The confocal grading of gastric intestinal metaplasia (CGGIM) may be used to assess a patient's risk by the endoscopic assessment of IM in the antrum, incisura, and corpus with the use of confocal laser endomicroscopy. The minimum score is 0 and the maximum score is 10. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients. CGGIM scores were calculated to be compared with OLGIM based on the results of the endoscopist 's procedure.
AI yielded the sensitivity of CGGIM score in the diagnosis of OLGIM III/IV | 2 years
  The confocal grading of gastric intestinal metaplasia (CGGIM) may be used to assess a patient's risk by the endoscopic assessment of IM in the antrum, incisura, and corpus with the use of confocal laser endomicroscopy. The minimum score is 0 and the maximum score is 10. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients. CGGIM scores were calculated based on existing AI model identification results and compared with OLGIM.
AI yielded the specificity of CGGIM score in the diagnosis of OLGIM III/IV | 2 years
  The confocal grading of gastric intestinal metaplasia (CGGIM) may be used to assess a patient's risk by the endoscopic assessment of IM in the antrum, incisura, and corpus with the use of confocal laser endomicroscopy. The minimum score is 0 and the maximum score is 10. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients. CGGIM scores were calculated based on existing AI model identification results and compared with OLGIM.
AI yields accuracy of CGGIM score for diagnosis of OLGIM III/IV | 2 years
  The confocal grading of gastric intestinal metaplasia (CGGIM) may be used to assess a patient's risk by the endoscopic assessment of IM in the antrum, incisura, and corpus with the use of confocal laser endomicroscopy. The minimum score is 0 and the maximum score is 10. The higher the score, the more severe the degree of intestinal metaplasia, and the higher the risk of gastric cancer in patients. CGGIM scores were calculated based on existing AI model identification results and compared with OLGIM.

SECONDARY OUTCOMES:
Comparison of accuracy of CGGIM score between AI and endoscopists in diagnosing OLGIM III/IV | 2 years
  Chi-square test was used to compare the accuracy of endoscopists and AI in the diagnosis of OLGIM

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, QiLu Hospital, Shandong University, Jinan, Shandong, China